CLINICAL TRIAL: NCT01485614
Title: A Phase III, Multicenter, Double-Blind, Randomized, Placebo-Controlled Clinical Trial to Evaluate the Safety and Efficacy of Sitagliptin in Pediatric Patients With Type 2 Diabetes Mellitus With Inadequate Glycemic Control
Brief Title: Study to Assess Safety & Efficacy of Sitagliptin as Initial Oral Therapy for Treatment of Type 2 Diabetes Mellitus in Pediatric Participants. (MK-0431-083)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-083; 2011-002528-42 (EudraCT Number); MK-0431-083 (Other: Merck Protocol Number)
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sitagliptin (Experimental): Participants will receive 1 tablet of sitagliptin 100 mg prior to the morning meal and 2 tablets of placebo matching metformin 500 mg prior to both the morning and evening meals during Weeks 0-20. Participants will continue to receive 1 tablet of sitagliptin 100 mg prior to the morning meal and 2 tablets of placebo matching metformin 500 mg prior to both the morning and evening meals during Weeks 20-54.
  Interventions: Drug: Sitagliptin; Drug: Placebo to metformin; Drug: Glycemic Rescue 1; Biological: Glycemic Rescue 2
- Placebo/Metformin (Placebo Comparator): Participants will receive 1 tablet of placebo matching sitagliptin 100 mg prior to the morning meal and 2 tablets of placebo matching metformin 500 mg prior to both the morning and evening meals during Weeks 0-20. Participants will receive 1 tablet of placebo matching sitagliptin 100 mg prior to the morning meal and 2 tablets of metformin 500 mg prior to both the morning and evening meals during Weeks 20-54.
  Interventions: Drug: Metformin; Drug: Placebo to sitagliptin; Drug: Placebo to metformin; Drug: Glycemic Rescue 1; Biological: Glycemic Rescue 2
- Metformin (Active Comparator): Participants will receive 1 tablet of placebo matching sitagliptin 100 mg prior to the morning meal and 2 tablets of metformin 500 mg prior to both the morning and evening meals during Weeks 0-20. Participants will continue to receive 1 tablet of placebo matching sitagliptin 100 mg prior to the morning meal and 2 tablets of metformin 500 mg prior to both the morning and evening meals during Weeks 20-54.
  Interventions: Drug: Metformin
- Placebo/Sitagliptin (Placebo Comparator): Participants will receive 1 tablet of placebo matching sitagliptin 100 mg prior to the morning meal and 2 tablets of placebo matching metformin 500 mg prior to both the morning and evening meals during Weeks 0-20. Participants will receive 1 tablet of sitagliptin 100 mg prior to the morning meal and 2 tablets of placebo matching metformin 500 mg prior to both the morning and evening meals during Weeks 20-54.
  Interventions: Drug: Sitagliptin; Drug: Placebo to sitagliptin; Drug: Placebo to metformin

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100 mg tablet administered orally once daily
  Other Names: Januvia®, Tesavel®, Xelevia®, Ristaben®, Glactiv®
  Arms: Placebo/Sitagliptin; Sitagliptin
Drug: Metformin — Metformin 500 mg tablets administered orally starting at 500 mg/day and uptitrated by 500 mg every week to a final dose of 1000 mg twice daily
  Other Names: Glucophage®, Metgluco®, Glycoran®
  Arms: Metformin; Placebo/Metformin
Drug: Placebo to sitagliptin — Matching placebo to sitagliptin 100 mg tablet administered orally once daily
  Arms: Placebo/Metformin; Placebo/Sitagliptin
Drug: Placebo to metformin — Matching placebo to metformin 500 mg tablets, 2 tablets administered orally twice daily
  Arms: Placebo/Metformin; Placebo/Sitagliptin; Sitagliptin
Drug: Glycemic Rescue 1 — Participants in the sitagliptin arm who require glycemic rescue will receive metformin during Weeks 0-20 and Weeks 20-54. Participants in the placebo arm who require glycemic rescue will receive metformin during Weeks 0-20. Participants in the placebo arm who have switched to metformin during Weeks 20-54 and require glycemic rescue will receive sitagliptin.
  Arms: Placebo/Metformin; Sitagliptin
Biological: Glycemic Rescue 2 — Participants who require glycemic rescue after Glycemic Rescue 1 will receive open-label insulin. Participants on background insulin therapy will have the dose of their background insulin up-titrated.
  Arms: Placebo/Metformin; Sitagliptin

SUMMARY:
The purpose of the study is to assess the safety of the addition of sitagliptin, and its effect on hemoglobin A1c (A1C) in pediatric participants 10-17 years of age with type 2 diabetes mellitus (T2DM) with inadequate glycemic control. The primary hypothesis for this study is that sitagliptin reduces A1C more than placebo after 20 weeks of treatment.

DETAILED DESCRIPTION:
This trial is of approximately 56 weeks in duration, including a screening period of up to 1 week, a 1-week single-blind placebo run-in period, a 20-week placebo-controlled, double blind treatment period [Phase A] and a 34-week double-blind active controlled treatment period [Phase B] during which participants randomized to the placebo arm who have not initiated glycemic rescue therapy with metformin during Phase A will receive metformin (in a blinded manner). A telephone contact will be performed 14 days after the last dose of study medication to assess for any serious adverse events (SAEs).

Participants enrolled in the metformin and placebo/sitagliptin arms prior to implementation of Protocol Amendment 05 completed the study on their original treatment assignments.

EUPASS4468 is a follow-up, non-interventional, observational assessment of safety of participants who participated in the MK-0431-083 study for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus (T2DM)
* Has not received treatment with an antihyperglycemic agent (AHA) for ≥12 weeks prior to the Screening Visit/Visit 1, or is on a stable dose of insulin (without any other AHA) for at least 12 weeks prior to the Screening Visit/Visit 1. At screening, participants on insulin doses that are not stable can have their insulin doses adjusted and be eligible to participate after their dose remains stable for ≥12 weeks, if they meet all other eligibility criteria. In India, only participants on stable doses of insulin will be eligible.
* An A1C of ≥6.5% and ≤10.0% (For participants on insulin: an A1C ≥7.0% and ≤10.0%).

Exclusion Criteria:

* History of type 1 diabetes mellitus, autoimmune diabetes mellitus or has a positive antibody screen for anti-GAD (Glutamic Acid Decarboxylase) or (Islet cell autoantigen) ICA-512.
* Known monogenic diabetes, secondary diabetes, or a genetic syndrome or disorder known to affect glucose tolerance other than diabetes.
* Symptomatic hyperglycemia and/or moderate to large ketonuria and/or positive test for ketonemia requiring immediate initiation of antihyperglycemic therapy.
* Previously taken a DPP-4 (Dipeptidyl peptidase-4) inhibitor (such as sitagliptin, vildagliptin, alogliptin, or saxagliptin) or GLP-1 (Glucagon-like peptide-1) receptor agonist (such as exenatide or liraglutide).
* Hypersensitivity or contraindication (according to the product circular in the country of the investigational site) to metformin.
* Chronic treatment with a medication known to cause weight gain within 30 days of study start or weight loss or increased blood glucose within 8 weeks of study start or treated with an anti-psychotic within the past 12 weeks.
* On a weight loss program and not in the maintenance phase or have undergone bariatric surgery within 12 months prior to study start.
* On or likely to require treatment with ≥14 consecutive days or repeated courses of pharmacologic doses of corticosteroids.
* Undergone a surgical procedure within the prior 4 weeks or has major surgery planned during the study.
* History of congenital heart disease or cardiovascular disease other than hypertension.
* Medical history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease.
* Active nephropathy (i.e., nephrotic syndrome or glomerulonephritis).
* Chronic myopathy, mitochondrial disorder, or a progressive neurological or neuromuscular disorder (e.g., polymyositis, or multiple sclerosis).
* Human immunodeficiency virus (HIV) as assessed by medical history.
* Clinically significant hematological disorder (such as aplastic anemia, thrombocytopenia, myeloproliferative or myelodysplastic syndrome).
* Under treatment for hyperthyroidism.
* Exhibits abnormal growth patterns or is being treated with growth hormone.
* History of malignancy or clinically important hematologic disorder.
* History of idiopathic acute pancreatitis or chronic pancreatitis.
* Known history of recreational or illicit drug use, or of alcohol abuse or dependence (within the past year).
* Donated blood products or has had phlebotomy of >10% of estimated total blood volume within 8 weeks of signing informed consent, or intends to donate blood products or receive blood products within the projected duration of the study.
* Pregnant, has a positive urine pregnancy test at Screening Visit/Visit 1, is expecting to conceive within the projected duration of the study, or is breast-feeding.
* Exclusionary laboratory values.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2012-02-10 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Shankar RR, Zeitler P, Deeb A, Jalaludin MY, Garcia R, Newfield RS, Samoilova Y, Rosario CA, Shehadeh N, Saha CK, Zhang Y, Zilli M, Scherer LW, Lam RLH, Golm GT, Engel SS, Kaufman KD. A randomized clinical trial of the efficacy and safety of sitagliptin as initial oral therapy in youth with type 2 diabetes. Pediatr Diabetes. 2022 Mar;23(2):173-182. doi: 10.1111/pedi.13279. Epub 2021 Dec 22. PMID 34779087

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited participants in clinics/clinical offices in 42 countries.
Pre-assignment Details: Participants in a one-week, run-in received sitagliptin placebo prior to morning meals and metformin placebo prior to morning and evening meals.
  Participants enrolled in the metformin and placebo/sitagliptin arms prior to implementation of Protocol Amendment 05 completed the study on their original treatment assignments.
Groups:
- Sitagliptin: Participants received 1 tablet of sitagliptin 100 mg prior to the morning meal and 2 tablets of placebo matching metformin 500 mg prior to both the morning and evening meals during Weeks 0-20. Participants continued to receive 1 tablet of sitagliptin 100 mg prior to the morning meal and 2 tablets of placebo matching metformin 500 mg prior to both the morning and evening meals during Weeks 20-54.
- Placebo/Metformin: Participants received 1 tablet of placebo matching sitagliptin 100 mg prior to the morning meal and 2 tablets of placebo matching metformin 500 mg prior to both the morning and evening meals during Weeks 0-20. Participants received 1 tablet of placebo matching sitagliptin 100 mg prior to the morning meal and 2 tablets of metformin 500 mg prior to both the morning and evening meals during Weeks 20-54.
- Metformin: Participants received 1 tablet of placebo matching sitagliptin 100 mg prior to the morning meal and 2 tablets of metformin 500 mg prior to both the morning and evening meals during Weeks 0-20. Participants continued to receive 1 tablet of placebo matching sitagliptin 100 mg prior to the morning meal and 2 tablets of metformin 500 mg prior to both the morning and evening meals during Weeks 20-54.
- Placebo/Sitagliptin: Participants received 1 tablet of placebo matching sitagliptin 100 mg prior to the morning meal and 2 tablets of placebo matching metformin 500 mg prior to both the morning and evening meals during Weeks 0-20. Participants received 1 tablet of sitagliptin 100 mg prior to the morning meal and 2 tablets of placebo matching metformin 500 mg prior to both the morning and evening meals during Weeks 20-54.
Period: Randomization
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Started | 96 | 90 | 9 | 5
Completed | 95 | 90 | 9 | 5
Not Completed | 1 | 0 | 0 | 0
Not completed — Not Treated | 1 | 0 | 0 | 0
Period: Weeks 0-20
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Started | 95 | 90 | 9 | 5
Treated | 95 | 90 | 9 | 5
Completed | 85 | 86 | 8 | 5
Not Completed | 10 | 4 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 5 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 1 | 0
Period: Weeks 20-54
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Started | 85 | 86 | 8 | 5
Completed | 74 | 78 | 6 | 5
Not Completed | 11 | 8 | 2 | 0
Not completed — Lost to Follow-up | 4 | 3 | 1 | 0
Not completed — Withdrawal by Parent/Guardian | 2 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population consisted of all randomized and treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin | Total
Number analyzed (Participants) | 95 | 90 | 9 | 5 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (2.0) | 13.7 (1.9) | 13.3 (3.0) | 15.0 (1.6) | 14.0 (2.0)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0 | 0 | 0
  Children (2-11 years) | 11 | 11 | 3 | 0 | 25
  Adolescents (12-17 years) | 84 | 79 | 6 | 5 | 174
  Adults (18-64 years) | 0 | 0 | 0 | 0 | 0
  From 65-84 years | 0 | 0 | 0 | 0 | 0
  85 years and over | 0 | 0 | 0 | 0 | 0
  Unknown | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 58 | 6 | 3 | 121
  Male | 41 | 32 | 3 | 2 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 33 | 2 | 2 | 73
  Not Hispanic or Latino | 53 | 54 | 5 | 3 | 115
  Unknown or Not Reported | 6 | 3 | 2 | 0 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 9 | 0 | 0 | 15
  Asian | 13 | 14 | 1 | 2 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 2 | 1 | 0 | 11
  White | 48 | 47 | 6 | 3 | 104
  More than one race | 20 | 18 | 1 | 0 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Glycated Hemoglobin (A1C) [Mean (Standard Deviation); unit: Percentage] — A1C is a blood marker used to report average blood glucose levels over prolonged periods of time. A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. The analysis population includes all randomized participants who received ≥1 dose of study medication and had a baseline measurement of A1C.
  Percentage | 7.43 (1.02) | 7.56 (1.08) | 7.43 (1.07) | 8.02 (0.75) | 7.50 (1.04)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] — Blood glucose was measured on a fasting basis.
  mg/dL | 138.4 (47.2) | 138.6 (42.8) | 134.6 (59.1) | 142.2 (38.7) | 138.6 (44.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C (A1C) at Week 20
Description: Glycated hemoglobin (A1C) is a blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Change from baseline was estimated as the Week 20 A1C minus the Week 0 A1C.
Time Frame: Baseline and Week 20
Population: The analysis population included all randomized participants who received ≥1 dose of study medication and had data for the analysis endpoint at both baseline and Week 20.
Measure: Mean (Standard Deviation); unit: Percentage
Groups:
- Sitagliptin: Participants received 1 tablet of sitagliptin 100 mg prior to the morning meal and 2 tablets of placebo matching metformin 500 mg prior to both the morning and evening meals during Weeks 0-20.
- Placebo/Metformin; Placebo/Sitagliptin: Participants received 1 tablet of placebo matching sitagliptin 100 mg prior to the morning meal and 2 tablets of placebo matching metformin 500 mg prior to both the morning and evening meals during Weeks 0-20.
- Metformin: Participants received 1 tablet of placebo matching sitagliptin 100 mg prior to the morning meal and 2 tablets of metformin 500 mg prior to both the morning and evening meals during Weeks 0-20.
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 78 | 70 | 8 | 3
Percentage | -0.13 (1.58) [lower limit 1.58] | -0.02 (1.45) [lower limit 1.45] | -1.03 (0.72) [lower limit 0.72] | 0.57 (1.62) [lower limit 1.62]

2. Primary Outcome: Baseline Glycated Hemoglobin (A1C) for the Placebo (Pooled) Arm
Description: A1C is a blood marker used to report average blood glucose levels over prolonged periods of time. A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. The Placebo (pooled) arm was a pooling of the Placebo/Metformin and Placebo/Sitagliptin arms for analysis purposes.
Time Frame: Baseline
Population: The analysis population included all randomized participants who received ≥1 dose of study medication and had a baseline measurement of A1C.
Measure: Mean (Standard Deviation); unit: Percentage
Groups:
- Placebo (Pooled): Participants received placebo from Week 0-20.
Arm/Group | Placebo (Pooled)
Number analyzed (Participants) | 95
Percentage | 7.58 (1.06)

3. Primary Outcome: Change From Baseline In A1C at Week 20 (Analysis of Selected Arms: Sitagliptin and Placebo (Pooled))
Description: Glycated hemoglobin (A1C) is a blood marker used to report average blood glucose levels over time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Mean change from baseline was estimated as the Week 20 A1C minus the Week 0 A1C from a longitudinal data analysis (LDA) model. The placebo arm in this comparison is a pooling of the Placebo/Metformin and Placebo/Sitagliptin arms. The Statistical Analysis Plan (SAP) did not specify for the Metformin arm to be included in statistical comparisons, so results for this arm are provided separately.
Time Frame: Baseline and Week 20
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Sitagliptin | Placebo (Pooled)
Number analyzed (Participants) | 95 | 95
Percentage | -0.01 [-0.35 to 0.34] | 0.18 [-0.17 to 0.53]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo (Pooled); Test type: Superiority; p = 0.448, Mixed Models Analysis; The Least Squares (LS) Mean for the arm "Sitagliptin" is compared against that of "Placebo (pooled)"; Least Squares Means Difference = -0.19, 95% CI 2-sided [-0.68 to 0.30]

4. Primary Outcome: Number of Participants Who Experienced ≥1 Adverse Event During Weeks 0-56
Description: The number of participants experiencing ≥1 adverse event during Weeks 0-56 was reported. An adverse event is defined as any untoward medical occurrence in a person administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to Week 56
Population: The analysis population includes all randomized participants who received ≥1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 95 | 90 | 9 | 5
Participants | 73 | 67 | 7 | 4

5. Primary Outcome: Percentage of Participants Who Experienced ≥1 Adverse Event During Weeks 0-56 (Analysis of Selected Arms: Sitagliptin and Placebo/Metformin)
Description: The number of participants experiencing ≥1 adverse event during Weeks 0-56 was reported. An adverse event is any untoward medical occurrence in a person administered a pharmaceutical product and does not have to have a causal relationship with this treatment. The SAP did not specify for the Metformin arm to be included in statistical comparisons, so results for this arm are provided separately.
Time Frame: Up to Week 56
Population: The analysis population includes all randomized participants who received ≥1 dose of study medication. Participants (n=5) from the Placebo/Sitagliptin arm were excluded because sitagliptin received during Week 0-54 was an inappropriate control for the Sitagliptin arm which received sitagliptin during both study treatment phases.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo/Metformin
Number analyzed (Participants) | 95 | 90
Percentage of participants | 76.8 | 74.4
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo/Metformin; Test type: Other; Percentage of participants with ≥1 adverse event for the arm "Sitagliptin" was compared against that of "Placebo/Metformin" with Miettinen & Nurminen; Difference in Percentage = 2.4, 95% CI 2-sided [-10.0 to 14.9]

6. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event During Weeks 0-54
Description: The number of participants who discontinued from study drug due to an adverse event during Weeks 0-54 was reported. An adverse event is defined as any untoward medical occurrence in a person administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to Week 54
Population: The analysis population includes all randomized participants who received ≥1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 95 | 90 | 9 | 5
Participants | 5 | 1 | 0 | 0

7. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event During Weeks 0-54 (Analysis of Selected Arms: Sitagliptin and Placebo/Metformin)
Description: The percentage of participants who discontinued from study drug due to an adverse event during Weeks 0-54 was reported. An adverse event is any untoward medical occurrence in a person administered a pharmaceutical product and does not have to have a causal relationship with this treatment. The SAP did not specify for the Metformin arm to be included in statistical comparisons, so results for this arm are provided separately.
Time Frame: Up to Week 54
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo/Metformin
Number analyzed (Participants) | 95 | 90
Percentage of participants | 5.3 | 1.1
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo/Metformin; Test type: Other; [p-value comment as in outcome 5, analysis 1]; Difference in percentage = 4.2, 95% CI 2-sided [-1.3 to 10.8]

8. Secondary Outcome: Change From Baseline in A1C at Week 54
Description: A1C is a blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. This change from baseline reflects the Week 54 A1C minus the Week 0 A1C.
Time Frame: Baseline and Week 54
Population: The analysis population included all randomized participants who took at least one dose of study medication and had data for the analysis endpoint at both baseline and Week 54.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 41 | 48 | 4 | 1
Percentage | -0.19 (1.37) | -0.90 (1.41) | -0.70 (0.94) | -0.50 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

9. Secondary Outcome: Percentage of Participants With A1C at Goal (<7.0%) at Week 20
Description: The percentage of participants with A1C at goal (<7.0%) at Week 20 was presented. All numbers shown in each individual treatment arm are based on the observed values (Missing = Not at Goal).
Time Frame: Week 20
Population: The analysis population included all randomized participants who received ≥1 dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 95 | 90 | 9 | 5
Percentage of Participants | 49.5 | 37.8 | 77.8 | 20.0

10. Secondary Outcome: Percentage of Participants With A1C at Goal (<7.0%) at Week 20 (Analysis of Selected Arms: Sitagliptin and Placebo (Pooled))
Description: The percentage of participants with A1C at goal (<7.0%) at Week 20 was presented. The analysis table includes the observed values for each treatment arm (Missing = Not at Goal) and the estimated treatment difference (Missing = Multiple Imputation). The current outcome measure focused on comparing results from participants randomized to sitagliptin or placebo. The Placebo arm in this comparison was a pooling of the Placebo/Metformin and Placebo/Sitagliptin arms. The SAP did not specify for the Metformin arm to be included in statistical comparisons, so results for this arm are provided separately.
Time Frame: Week 20
Population: The analysis population included all randomized participants who received ≥1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo (Pooled)
Number analyzed (Participants) | 95 | 95
Percentage of participants | 49.5 | 36.8
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo (Pooled); Test type: Superiority; p = 0.374, Miettinen and Nurminen — Percentage of participants with an A1C goal (7.0%) in the arm "Sitagliptin" was compared against the arm "Placebo (pooled)"; Difference in percentage = 6.7, 95% CI 2-sided [-8.1 to 21.2]; For estimating the treatment difference, when the A1C result for a participant at Week 20 was not available, a multiple imputation method based on the Linear Discriminant Analysis (LDA) model was used to impute whether the participant had met the goal

11. Secondary Outcome: Percentage of Participants With A1C at Goal (<6.5%) at Week 20
Description: The percentage of participants with A1C at goal (<6.5%) at Week 20 was presented. All numbers shown in each individual treatment arm are based on the observed values (Missing = Not at Goal).
Time Frame: Week 20
Population: The analysis population included all randomized participants who received ≥1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 95 | 90 | 9 | 5
Percentage of participants | 30.5 | 23.3 | 66.7 | 20.0

12. Secondary Outcome: Percentage of Participants With A1C at Goal (<6.5%) at Week 20 (Analysis of Selected Arms: Sitagliptin and Placebo (Pooled))
Description: The percentage of participants with A1C at goal (<6.5%) at Week 20 was presented. The analysis table includes the observed values for each treatment arm (Missing = Not at Goal) and the estimated treatment difference (Missing = Multiple Imputation). The current outcome measure focused on comparing results from participants randomized to sitagliptin or placebo. The Placebo arm in this comparison was a pooling of the Placebo/Metformin and Placebo/Sitagliptin arms. The SAP did not specify for the Metformin arm to be included in statistical comparisons, so results for this arm are provided separately.
Time Frame: Week 20
Population: The analysis population included all randomized participants who received ≥1 dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sitagliptin | Placebo (Pooled)
Number analyzed (Participants) | 95 | 95
Percentage of Participants | 30.5 | 23.2
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo (Pooled); Test type: Superiority; p = 0.639, Miettinen and Nurminen; The percentage of participants with an A1C at the A1C goal (6.5%) in the arm "Sitagliptin" was compared against the arm "Placebo (pooled)"; Difference in percentage = 3.6, 95% CI 2-sided [-11.6 to 18.3]; For estimating the treatment difference, when the A1C result for a participant at Week 20 was not available, a multiple imputation method based on the LDA model was used to impute whether the participant had met the goal

13. Secondary Outcome: Percentage of Participants With A1C at Goal (<7.0%) at Week 54
Description: The percentage of participants with A1C at goal (<7.0%) at Week 54 was presented. All numbers shown in each individual treatment arm are based on the observed values (Missing = Not at Goal).
Time Frame: Week 54
Population: The analysis population included all randomized participants who received ≥1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 95 | 90 | 9 | 5
Percentage of participants | 28.4 | 40.0 | 33.3 | 20.0

14. Secondary Outcome: Percentage of Participants With A1C at Goal (<6.5%) at Week 54
Description: The percentage of participants with A1C at goal (<6.5%) at Week 54 was presented. All numbers shown in each individual treatment arm are based on the observed values (Missing = Not at Goal).
Time Frame: Week 54
Population: The analysis population included all randomized participants who received ≥1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 95 | 90 | 9 | 5
Percentage of participants | 20.0 | 35.6 | 22.2 | 20.0

15. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 20
Description: Blood glucose was measured on a fasting basis. Change in plasma glucose levels was FPG at Week 20 minus FPG at baseline.
Time Frame: Baseline and Week 20
Population: The analysis population included all randomized participants who received ≥1 dose of study medication and had data for the analysis endpoint both at baseline and Week 20.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 81 | 74 | 8 | 3
mg/dL | 9.98 (61.86) [lower limit 61.86] | 7.59 (41.11) [lower limit 41.11] | -19.88 (49.78) [lower limit 49.78] | 57.67 (51.05) [lower limit 51.05]

16. Secondary Outcome: Baseline Fasting Plasma Glucose (FPG) for the Placebo (Pooled) Arm
Description: Blood glucose was measured on a fasting basis. The Placebo (pooled) arm was a pooling of the Placebo/Metformin and Placebo/Sitagliptin arms for analysis purposes.
Time Frame: Baseline
Population: The analysis population included all randomized participants who received ≥1 dose of study medication and had data for the analysis endpoint at baseline.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo (Pooled)
Number analyzed (Participants) | 95
mg/dL | 138.8 (42.4)

17. Secondary Outcome: Change From Baseline in FPG at Week 20 (Analysis of Selected Arms: Sitagliptin and Placebo (Pooled))
Description: Blood glucose was measured on a fasting basis. Change in plasma glucose levels was FPG at Week 20 minus FPG at baseline and was estimated from a longitudinal data analysis model. The current outcome measure focused on results from participants randomized to sitagliptin or placebo. The Week 20 treatment comparison of Sitagliptin vs Placebo included all participants treated with Sitagliptin or Placebo. The Placebo arm in this comparison was a pooling of the Placebo/Metformin and Placebo/Sitagliptin arms. The SAP did not specify for the Metformin arm to be included in statistical comparisons, so results for this arm are provided separately.
Time Frame: Baseline and Week 20
Population: The analysis population includes all randomized participants who received ≥1 dose of study medication and had data for the analysis endpoint at both baseline and Week 20.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo (Pooled)
Number analyzed (Participants) | 95 | 95
mg/dL | 7.2 [-4.2 to 18.7] | 5.7 [-6.0 to 17.4]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo (Pooled); Test type: Superiority; p = 0.849, Mixed Models Analysis; The Least Squares (LS) Mean for the arm "Sitagliptin" was compared against that of "Placebo (pooled)"; Least Squares Means Difference = 1.5, 95% CI 2-sided [-14.4 to 17.5]

18. Secondary Outcome: Change From Baseline in FPG at Week 54
Description: Blood glucose was measured on a fasting basis. Change in plasma glucose levels was FPG at Week 54 minus FPG at baseline.
Time Frame: Baseline and Week 54
Population: The analysis population included all randomized participants who received ≥1 dose of study medication and had data for the analysis endpoint both at baseline and Week 54.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 44 | 51 | 6 | 1
mg/dL | -3.03 (48.55) | -4.52 (50.68) | -29.92 (53.19) | 3.00 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

19. Secondary Outcome: Change From Baseline in 2-Hour Post-meal Glucose (PMG) at Week 20
Description: PMG endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. This change from baseline was Week 20 2-hour PMG minus the Week 0 2-hour PMG.
Time Frame: Baseline and Week 20
Population: The analysis population included all randomized participants who received ≥1 dose of study medication, consented to participate in the MTT, and had data for the analysis endpoint both at baseline and Week 20.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 12 | 12 | 4 | 2
mg/dL | -2.9 (42.6) [lower limit 42.6] | 2.1 (72.1) [lower limit 72.1] | -6.8 (21.1) [lower limit 21.1] | 63.5 (171.8) [lower limit 171.8]

20. Secondary Outcome: Change From Baseline in 2-hour PMG at Week 54
Description: PMG endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. This change from baseline was Week 54 2-hour PMG minus the Week 0 2-hour PMG.
Time Frame: Baseline and Week 54
Population: The analysis population included all randomized participants who received ≥1 dose of study medication, consented to participate in the MTT, and had data for the analysis endpoint both at baseline and Week 54.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 7 | 8 | 3 | 1
mg/dL | -1.7 (21.3) | -16.8 (48.9) | -39.7 (32.3) | -28.0 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

21. Secondary Outcome: Change From Baseline in 2-hour Incremental PMG at Week 20
Description: 2-Hour incremental PMG = Glucose at 120 minutes - glucose at 0 minutes. PMG endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. This change from baseline was Week 20 2-hour incremental PMG minus the Week 0 2-hour incremental PMG.
Time Frame: Baseline and Week 20
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 12 | 12 | 4 | 2
mg/dL | 1.5 (55.3) [lower limit 55.3] | 0.7 (35.9) [lower limit 35.9] | 0.8 (15.6) [lower limit 15.6] | 12.5 (98.3) [lower limit 98.3]

22. Secondary Outcome: Change From Baseline in 2-Hour Incremental PMG at Week 54
Description: 2-Hour incremental PMG = Glucose at 120 minutes - glucose at 0 minutes. PMG endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. This change from baseline was Week 54 2-hour incremental PMG minus the Week 0 2-hour incremental PMG.
Time Frame: Baseline and Week 54
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 7 | 8 | 3 | 1
mg/dL | -0.6 (64.6) | -26.6 (39.0) | -31.3 (34.8) | -32.0 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

23. Secondary Outcome: Change From Baseline in Insulin at Week 20 for Participants Not on Background Insulin
Description: This change from baseline reflects the Week 20 insulin minus the Week 0 insulin.
Time Frame: Baseline and Week 20
Population: The analysis population included all randomized participants not on background insulin who received ≥1 dose of study medication and had data for the analysis endpoint at both baseline and Week 20.
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 67 | 58 | 7 | 3
mIU/L | 1.59 (47.24) [lower limit 47.24] | -3.91 (22.31) [lower limit 22.31] | -7.25 (60.58) [lower limit 60.58] | -1.23 (20.55) [lower limit 20.55]

24. Secondary Outcome: Change From Baseline in Insulin at Week 54 For Participants Not on Background Insulin
Description: This change from baseline reflects the Week 54 insulin minus the Week 0 insulin.
Time Frame: Baseline and Week 54
Population: The analysis population included all randomized participants not on background insulin who received ≥1 dose of study medication and had data for the analysis endpoint both at baseline and Week 54.
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 37 | 45 | 5 | 1
mIU/L | -9.65 (40.82) | -6.64 (32.01) | -20.50 (65.08) | -9.95 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

25. Secondary Outcome: Change From Baseline in Proinsulin at Week 20 For Participants Not on Background Insulin
Description: This change from baseline reflects the Week 20 proinsulin minus the Week 0 proinsulin.
Time Frame: Baseline and Week 20
Population: The analysis population included all randomized participants not on background insulin who received ≥1 dose of study medication and had data for the analysis endpoint both at baseline and Week 20.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 68 | 57 | 7 | 3
pmol/L | 0.91 (81.88) [lower limit 81.88] | -10.88 (55.12) [lower limit 55.12] | 12.57 (36.98) [lower limit 36.98] | -1.33 (9.07) [lower limit 9.07]

26. Secondary Outcome: Change From Baseline in Proinsulin at Week 54 For Participants Not on Background Insulin
Description: This change from baseline reflects the Week 54 proinsulin minus the Week 0 proinsulin.
Time Frame: Baseline and Week 54
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 38 | 42 | 5 | 1
pmol/L | -10.62 (67.54) | -16.13 (81.52) | -23.30 (42.36) | -0.50 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

27. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio at Week 20 for Participants Not on Background Insulin
Description: Change from baseline was the Week 20 proinsulin/insulin ratio minus the Week 0 proinsulin/insulin ratio.
Time Frame: Baseline and Week 20
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 65 | 55 | 6 | 3
Ratio | 0.02 (0.22) [lower limit 0.22] | 0.02 (0.16) [lower limit 0.16] | -0.03 (0.10) [lower limit 0.10] | -0.19 (0.45) [lower limit 0.45]

28. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio at Week 54 For Participants Not on Background Insulin
Description: The change from baseline was Week 54 proinsulin/insulin ratio minus the Week 0 proinsulin/insulin ratio.
Time Frame: Baseline and Week 54
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 36 | 41 | 5 | 1
Ratio | 0.02 (0.23) | -0.03 (0.19) | -0.01 (0.06) | 0.02 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

29. Secondary Outcome: Change From Baseline in Homeostatic Model Assessment of β-cell Function (HOMA-β) at Week 20 For Participants Not on Background Insulin
Description: HOMA-β = 20 × fasting insulin (in mcIU/mL) ÷ {[FPG (in mg/dL)/18] - 3.5}. The change from baseline was Week 20 HOMA-β minus the Week 0 HOMA-β.
Time Frame: Baseline and Week 20
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Percentage of Beta Cell Function
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 67 | 58 | 7 | 3
Percentage of Beta Cell Function | 15.72 (162.47) [lower limit 162.47] | -53.23 (296.23) [lower limit 296.23] | -1757.50 (4765.46) [lower limit 4765.46] | -64.78 (126.65) [lower limit 126.65]

30. Secondary Outcome: Change From Baseline in HOMA-β at Week 54 For Participants Not on Background Insulin
Description: HOMA-β = 20 × fasting insulin (in mcIU/mL) ÷ {[FPG (in mg/dL)/18] - 3.5}. This change from baseline was Week 54 HOMA-β minus the Week 0 HOMA-β.
Time Frame: Baseline and Week 54
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Percentage of Beta Cell Function
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 36 | 45 | 5 | 1
Percentage of Beta Cell Function | -41.15 (183.17) | -63.88 (339.74) | -1860.69 (4099.22) | -121.48 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

31. Secondary Outcome: Change From Baseline in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) at Week 20 For Participants Not on Background Insulin
Description: HOMA-IR = fasting insulin (in mcIU/mL) × FPG (in mg/dL) / (22.5×18). This change from baseline was Week 20 HOMA-IR minus the Week 0 HOMA-IR.
Time Frame: Baseline and Week 20
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Index of insulin resistance
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 67 | 58 | 7 | 3
Index of insulin resistance | -0.50 (31.62) [lower limit 31.62] | -0.86 (9.02) [lower limit 9.02] | -4.46 (34.65) [lower limit 34.65] | 2.58 (9.30) [lower limit 9.30]

32. Secondary Outcome: Change From Baseline in HOMA-IR at Week 54 For Participants Not on Background Insulin
Description: HOMA-IR = fasting insulin (in mcIU/mL) × FPG (in mg/dL) / (22.5×18). This change from baseline was Week 54 HOMA-IR minus the Week 0 HOMA-IR.
Time Frame: Baseline and Week 54
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Index of insulin resistance
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 36 | 45 | 5 | 1
Index of insulin resistance | -6.13 (34.86) | -1.30 (15.31) | -15.18 (36.41) | -2.21 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

33. Secondary Outcome: Change From Baseline in Glucose 3-Hour Total Area Under the Curve (AUC) at Week 20
Description: AUC endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. This change from baseline was Week 20 glucose 3-hour AUC minus the Week 0 glucose 3-hour AUC.
Time Frame: Baseline and Week 20 (-10 min. before ingesting the meal, 0 min. prior to the meal, 10, 20, 30, 60, 90, 120, 180 minutes after ingesting the meal)
Population: The analysis population included all randomized participants who received ≥1 dose of study medication, consented to participate in the MTT, and had data for the analysis endpoint at baseline and Week 20.
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 12 | 12 | 4 | 2
mg*hr/dL | -49.3 (103.6) [lower limit 103.6] | 2.0 (190.0) [lower limit 190.0] | 18.6 (50.9) [lower limit 50.9] | 191.0 (434.2) [lower limit 434.2]

34. Secondary Outcome: Change From Baseline in Insulin 3-hour AUC at Week 20
Description: AUC endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. This change from baseline was Week 20 insulin 3-hour AUC minus the Week 0 insulin 3-hour AUC.
Time Frame: as for outcome 33
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: µIU*hr/mL
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 12 | 12 | 2 | 2
µIU*hr/mL | -14.5 (128.0) [lower limit 128.0] | -32.8 (99.9) [lower limit 99.9] | 141.7 (206.1) [lower limit 206.1] | -145.6 (180.6) [lower limit 180.6]

35. Secondary Outcome: Change From Baseline in C-peptide 3-Hour AUC at Week 20
Description: AUC endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. This change from baseline was Week 20 C-peptide 3-hour AUC minus the Week 0 C-peptide 3-hour AUC.
Time Frame: as for outcome 33
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 12 | 12 | 2 | 2
ng*hr/mL | -1.8 (4.9) [lower limit 4.9] | -0.1 (3.3) [lower limit 3.3] | 5.9 (7.6) [lower limit 7.6] | -6.4 (7.1) [lower limit 7.1]

36. Secondary Outcome: Change From Baseline in Insulin 3-Hour AUC/ Glucose 3-Hour AUC Ratio at Week 20
Description: AUC endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. This change from baseline was Week 20 insulin total AUC/glucose total AUC ratio minus the Week 0 insulin total AUC/glucose total AUC ratio.
Time Frame: as for outcome 33
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: [µIU*hr/mL]/[mg*hr/dL]
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 12 | 12 | 2 | 2
[µIU*hr/mL]/[mg*hr/dL] | 0.0 (0.3) [lower limit 0.3] | -0.1 (0.3) [lower limit 0.3] | 0.2 (0.4) [lower limit 0.4] | -0.2 (0.3) [lower limit 0.3]

37. Secondary Outcome: Change From Baseline in Glucose Excursion 3-Hour AUC at Week 20
Description: AUC endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. Excursion AUC = Incremental AUC above the level at the start of the meal. AUC below the level at the start of the meal did not contribute to the Excursion AUC. This change from baseline was Week 20 glucose Excursion 3-hour AUC minus the Week 0 glucose Excursion 3-hour AUC.
Time Frame: as for outcome 33
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 12 | 12 | 4 | 2
mg*hr/dL | -43.5 (97.4) [lower limit 97.4] | 10.8 (58.6) [lower limit 58.6] | 39.8 (50.1) [lower limit 50.1] | 46.2 (201.9) [lower limit 201.9]

38. Secondary Outcome: Change From Baseline in Insulin Excursion 3-Hour AUC at Week 20
Description: AUC endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. Excursion AUC = Incremental AUC above the level at the start of the meal. AUC below the level at the start of the meal did not contribute to the Excursion AUC. This change from baseline was Week 20 insulin Excursion 3-hour AUC minus the Week 0 insulin Excursion 3-hour AUC.
Time Frame: as for outcome 33
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: µIU*hr/mL
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 12 | 12 | 2 | 2
µIU*hr/mL | -12.4 (89.4) [lower limit 89.4] | -19.4 (93.6) [lower limit 93.6] | 87.5 (124.5) [lower limit 124.5] | -82.8 (93.4) [lower limit 93.4]

39. Secondary Outcome: Change From Baseline in C-peptide Excursion 3-Hour AUC at Week 20
Description: AUC endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. Excursion AUC = Incremental AUC above the level at the start of the meal. AUC below the level at the start of the meal did not contribute to the Excursion AUC. This change from baseline was Week 20 C-peptide Excursion 3-hour AUC minus the Week 0 C-peptide Excursion 3-hour AUC.
Time Frame: as for outcome 33
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 12 | 12 | 2 | 2
ng*hr/ml | -1.1 (3.1) [lower limit 3.1] | -0.4 (4.4) [lower limit 4.4] | 4.1 (5.6) [lower limit 5.6] | -4.8 (5.2) [lower limit 5.2]

40. Secondary Outcome: Change From Baseline in Insulin Excursion 3-Hour AUC/Glucose Excursion 3-Hour AUC Ratio at Week 20
Description: AUC endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. Excursion AUC = Incremental AUC above the level at the start of the meal. AUC below the level at the start of the meal did not contribute to the Excursion AUC. This change from baseline was Week 20 insulin Excursion 3-hour AUC/glucose Excursion 3-hour AUC ratio minus the Week 0 insulin Excursion 3-hour AUC/glucose Excursion 3-hour AUC ratio.
Time Frame: as for outcome 33
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: [μIU*hr/mL]/[mg*hr/dL]
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 11 | 10 | 2 | 2
[μIU*hr/mL]/[mg*hr/dL] | 2.2 (9.6) [lower limit 9.6] | 7.2 (17.5) [lower limit 17.5] | -2.5 (3.2) [lower limit 3.2] | 1.4 (2.2) [lower limit 2.2]

41. Secondary Outcome: Change From Baseline in Glucose 3-Hour AUC at Week 54
Description: AUC endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. This change from baseline was Week 54 glucose 3-hour AUC minus the Week 0 glucose 3-hour AUC.
Time Frame: Baseline and Week 54 (-10 min. before ingesting the meal, 0 min. prior to the meal, 10, 20, 30, 60, 90, 120, 180 minutes after ingesting the meal)
Population: The analysis population included all randomized participants who received ≥1 dose of study medication, consented to participate in the MTT, and had data for the analysis endpoint at baseline and Week 54.
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 7 | 8 | 3 | 1
mg*hr/dL | -21.1 (47.7) | -36.0 (136.1) | -73.1 (95.8) | -63.3 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

42. Secondary Outcome: Change From Baseline in Insulin 3-Hour AUC at Week 54
Description: AUC endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. This change from baseline was Week 54 insulin 3-hour AUC minus the Week 0 insulin 3-hour AUC.
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: µIU*hr/mL
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 7 | 8 | 2 | 1
µIU*hr/mL | -43.2 (259.8) | -253.9 (282.7) | -37.8 (9.4) | -184.4 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

43. Secondary Outcome: Change From Baseline in C-peptide 3-Hour AUC at Week 54
Description: AUC endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. This change from baseline was Week 54 C-peptide 3-hour AUC minus the Week 0 C-peptide 3-hour AUC.
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 7 | 8 | 2 | 1
ng*hr/ml | -0.1 (5.7) | -6.1 (8.2) | 1.7 (1.0) | -8.9 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

44. Secondary Outcome: Change From Baseline in Insulin 3-Hour AUC/Glucose 3-Hour AUC Ratio at Week 54
Description: AUC endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. This change from baseline was Week 54 insulin 3-hour AUC/glucose 3-hour AUC ratio minus the Week 0 insulin 3-hour AUC/glucose 3-hour AUC ratio.
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: [μIU*hr/mL]/[mg*hr/dL]
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 7 | 8 | 2 | 1
[μIU*hr/mL]/[mg*hr/dL] | -0.1 (0.5) | -0.6 (0.8) | -0.0 (0.2) | -0.3 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

45. Secondary Outcome: Change From Baseline in Glucose Excursion 3-Hour AUC at Week 54
Description: AUC endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. Excursion AUC = Incremental AUC above the level at the start of the meal. AUC below the level at the start of the meal did not contribute to the Excursion AUC. This change from baseline was Week 54 glucose Excursion 3-hour AUC minus the Week 0 glucose Excursion 3-hour AUC.
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 7 | 8 | 3 | 1
mg*hr/dL | -30.7 (100.7) | -50.1 (79.5) | -49.0 (87.5) | -74.0 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

46. Secondary Outcome: Change From Baseline in Insulin Excursion 3-Hour AUC at Week 54
Description: AUC endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. Excursion AUC = Incremental AUC above the level at the start of the meal. AUC below the level at the start of the meal did not contribute to the Excursion AUC. This change from baseline was Week 54 insulin Excursion 3-hour AUC minus the Week 0 insulin Excursion 3-hour AUC.
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: µIU*hr/mL
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 7 | 8 | 2 | 1
µIU*hr/mL | -103.8 (151.0) | -198.5 (263.0) | -40.2 (11.5) | -116.6 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

47. Secondary Outcome: Change From Baseline in C-Peptide Excursion 3-Hour AUC at Week 54
Description: AUC endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. Excursion AUC = Incremental AUC above the level at the start of the meal. AUC below the level at the start of the meal did not contribute to the Excursion AUC. This change from baseline was Week 54 C-peptide Excursion 3-hour AUC minus the Week 0 C-peptide Excursion 3-hour AUC.
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 7 | 8 | 2 | 1
ng*hr/ml | -1.8 (3.0) | -5.2 (8.8) | 0.9 (0.5) | -5.9 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

48. Secondary Outcome: Change From Baseline in Insulin Excursion 3-Hour AUC/Glucose Excursion 3-Hour AUC Ratio at Week 54
Description: AUC endpoints were derived via the trapezoidal rule using 9-point Meal Tolerance Test (MTT) measurements. Excursion AUC = Incremental AUC above the level at the start of the meal. AUC below the level at the start of the meal did not contribute to the Excursion AUC. This change from baseline was Week 54 insulin Excursion 3-hour AUC/glucose Excursion 3-hour AUC ratio minus the Week 0 insulin Excursion 3-hour AUC/glucose Excursion 3-hour AUC ratio.
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: [µIU*hr/mL]/[mg*hr/dL]
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 7 | 6 | 2 | 1
[µIU*hr/mL]/[mg*hr/dL] | 4.1 (13.1) | 3.7 (5.6) | -2.7 (4.3) | 1.4 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

49. Secondary Outcome: Percentage of Participants Initiating Glycemic Rescue Therapy by Week 20
Description: The percentage of participants who initiated glycemic rescue therapy prior to Week 20 was reported.
Time Frame: Up to Week 20
Population: The analysis population included all randomized participants who received ≥1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 95 | 90 | 9 | 5
Percentage of participants | 5.3 | 11.1 | 0.0 | 40.0

50. Secondary Outcome: Percentage of Participants Initiating Glycemic Rescue Therapy by Week 54
Description: The percentage of participants who initiated glycemic rescue therapy prior to Week 54 was reported.
Time Frame: Up to Week 54
Population: The analysis population included all randomized participants who received ≥1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 95 | 90 | 9 | 5
Percentage of participants | 35.8 | 28.9 | 11.1 | 80.0

51. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Week 20
Description: This change from baseline was Week 20 BMI minus the Week 0 BMI.
Time Frame: Baseline and Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 84 | 82 | 8 | 5
kg/m^2 | 0.0 (2.2) [lower limit 2.2] | -0.7 (1.9) [lower limit 1.9] | -0.8 (1.4) [lower limit 1.4] | -1.7 (2.8) [lower limit 2.8]

52. Secondary Outcome: Change From Baseline in BMI at Week 54
Description: This change from baseline was Week 54 BMI minus the Week 0 BMI.
Time Frame: Baseline and Week 54
Population: The analysis population included all randomized participants who received ≥1 dose of study medication and had data for the analysis endpoint at both baseline and Week 54.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 72 | 73 | 6 | 5
kg/m^2 | -0.4 (2.9) | -1.0 (2.9) | -0.6 (1.3) | -0.3 (1.6)

53. Secondary Outcome: Mean Percent Change of Peripheral Blood Mononuclear Cells Expressing CD26 From Baseline at Week 20
Description: The percent change from baseline in CD26 = ([CD26 value at Week 20] - [baseline CD26 value]) ÷ baseline CD26 value × 100.
Time Frame: Baseline and Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 68 | 57 | 4 | 3
Percent Change | 4.06 (19.25) [lower limit 19.25] | -1.78 (17.18) [lower limit 17.18] | 4.89 (1.90) [lower limit 1.90] | 14.57 (15.46) [lower limit 15.46]

54. Secondary Outcome: Mean Percent Change of Peripheral Blood Mononuclear Cells Expressing CD26 From Baseline at Week 54
Description: The percent change from baseline in CD26 = ([CD26 value at Week 54] - [baseline CD26 value]) ÷ baseline CD26 value × 100.
Time Frame: Baseline and Week 54
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 56 | 55 | 5 | 3
Percent Change | 4.74 (17.18) | 4.27 (18.24) | 12.63 (13.02) | -5.30 (4.19)

55. Secondary Outcome: Change From Baseline in Calcitonin at Week 20 - Females
Description: Calcitonin, along with parathyroid hormone, is a hormone that regulates calcium and bone metabolism. This change from baseline was Week 20 calcitonin minus the Week 0 calcitonin.
Time Frame: Baseline and Week 20
Population: The analysis population included all female randomized participants who received ≥1 dose of study medication and had data for the analysis endpoint at both baseline and Week 20.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 43 | 46 | 4 | 2
ng/L | -0.1 (0.5) [lower limit 0.5] | -2.0 (11.7) [lower limit 11.7] | 0.0 (0.0) [lower limit 0.0] | 0.0 (0.0) [lower limit 0.0]

56. Secondary Outcome: Change From Baseline in Calcitonin at Week 54 - Females
Description: Calcitonin, along with parathyroid hormone, is a hormone that regulates calcium and bone metabolism. This change from baseline was Week 54 calcitonin minus the Week 0 calcitonin.
Time Frame: Baseline and Week 54
Population: The analysis population included all female randomized participants who received ≥1 dose of study medication and had data for the analysis endpoint at both baseline and Week 54.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 30 | 43 | 3 | 2
ng/L | -1.0 (0.6) | -1.9 (12.1) | 0.0 (0.0) | 0.3 (0.4)

57. Secondary Outcome: Change From Baseline in Calcitonin at Week 20 - Males
Description: as for outcome 55
Time Frame: Baseline and Week 20
Population: The analysis population included all male randomized participants who received ≥1 dose of study medication and had data for the analysis endpoint at both baseline and Week 20.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 35 | 25 | 2 | 2
ng/L | 0.2 (1.4) [lower limit 1.4] | -0.2 (0.6) [lower limit 0.6] | -1.6 (2.2) [lower limit 2.2] | 0.5 (0.6) [lower limit 0.6]

58. Secondary Outcome: Change From Baseline in Calcitonin at Week 54 - Males
Description: as for outcome 56
Time Frame: Baseline and Week 54
Population: The analysis population included all male randomized participants who received ≥1 dose of study medication and had data for the analysis endpoint at both baseline and Week 54.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 33 | 21 | 1 | 2
ng/L | 0.1 (1.1) | -0.3 (0.9) | 0.0 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed. | 1.4 (0.3)

59. Secondary Outcome: Change From Baseline in Urine N-terminal Cross-linking Telopeptide of Bone Collagen [u-NTx]/Creatinine Ratio at Week 20 - Females
Description: Urine N-terminal cross-linking telopeptide of bone collagen [u-NTx]/creatinine ratio is a biochemical marker of bone turnover/resorption. BCE = Bone Collagen Equivalents
Time Frame: Baseline and Week 20
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: nmol(BCE)/mmol(creatinine)
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 33 | 31 | 4 | 3
nmol(BCE)/mmol(creatinine) | -28.7 (120.9) [lower limit 120.9] | -41.2 (148.9) [lower limit 148.9] | -98.0 (153.0) [lower limit 153.0] | 12.7 (29.2) [lower limit 29.2]

60. Secondary Outcome: Change From Baseline u-NTx/Creatinine Ratio at Week 20 - Males
Description: as for outcome 59
Time Frame: Baseline and Week 20
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: nmol(BCE)/mmol(creatinine)
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 31 | 21 | 1 | 2
nmol(BCE)/mmol(creatinine) | -30.9 (167.2) | -69.8 (162.1) | 62.0 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed. | -29.0 (32.5)

61. Secondary Outcome: Change From Baseline in u-NTx/Creatinine Ratio at Week 54 - Females
Description: Urine N-terminal cross-linking telopeptide of bone collagen [u-NTx]/creatinine ratio is a biochemical marker of bone turnover/resorption. Bone Collagen Equivalents
Time Frame: Baseline and Week 54
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: nmol(BCE)/mmol(creatinine)
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 28 | 30 | 4 | 3
nmol(BCE)/mmol(creatinine) | -88.4 (102.6) | -61.2 (137.6) | -80.3 (208.5) | -17.0 (13.5)

62. Secondary Outcome: Change From Baseline in u-NTx/Creatinine Ratio at Week 54 - Males
Description: Urine N-terminal cross-linking telopeptide of bone collagen [u-NTx]/creatinine ratio is a biochemical marker of bone turnover/resorption. All participants in the Metformin arm were missing baseline or Week 54 measurements. BCE = Bone Collagen Equivalents
Time Frame: Baseline and Week 54
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: nmol(BCE)/mmol(creatinine)
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 30 | 16 | 0 | 1
nmol(BCE)/mmol(creatinine) | -78.2 (166.9) | -102.4 (267.7) |  | -30.0 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

63. Secondary Outcome: Change From Baseline in Bone-Specific Alkaline Phosphatase at Week 20 - Females
Description: Bone-specific alkaline phosphatase is a biochemical marker of bone turnover. This change from baseline was Week 20 bone-specific alkaline phosphatase minus the Week 0 bone-specific alkaline phosphatase.
Time Frame: Baseline and Week 20
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 43 | 52 | 5 | 3
μg/L | -6.0 (13.7) [lower limit 13.7] | -4.2 (9.9) [lower limit 9.9] | -9.7 (7.7) [lower limit 7.7] | 10.7 (9.7) [lower limit 9.7]

64. Secondary Outcome: Change From Baseline in Bone-Specific Alkaline Phosphatase at Week 54 - Females
Description: Bone-specific alkaline phosphatase is a biochemical marker of bone turnover. This change from baseline was Week 54 bone-specific alkaline phosphatase minus the Week 0 bone-specific alkaline phosphatase.
Time Frame: Baseline and Week 54
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 30 | 43 | 4 | 3
μg/L | -20.0 (28.4) | -13.5 (18.1) | -14.9 (10.3) | -6.9 (9.2)

65. Secondary Outcome: Change From Baseline in Bone-Specific Alkaline Phosphatase at Week 20 - Males
Description: as for outcome 63
Time Frame: Baseline and Week 20
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 36 | 25 | 2 | 2
μg/L | -2.2 (21.6) [lower limit 21.6] | 0.1 (19.9) [lower limit 19.9] | -7.1 (0.2) [lower limit 0.2] | 4.7 (8.2) [lower limit 8.2]

66. Secondary Outcome: Change From Baseline in Bone-Specific Alkaline Phosphatase at Week 54 - Males
Description: as for outcome 64
Time Frame: Baseline and Week 54
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 33 | 20 | 1 | 2
μg/L | -16.2 (28.0) | -15.0 (27.0) | -1.3 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed. | -15.3 (12.4)

67. Secondary Outcome: Percent Change From Baseline in Insulin-like Growth Factor-1 (IGF-1) at Week 20 - Females
Description: IGF-1 is a biochemical marker of growth hormone action and growth. The percent change from baseline in IGF-1 = ([IGF-1 value at Week 20] - [baseline IGF-1 value]) ÷ [baseline IGF-1 value] × 100.
Time Frame: Baseline and Week 20
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 38 | 49 | 5 | 2
Percent Change | 0.5 (21.9) [lower limit 21.9] | 11.0 (34.0) [lower limit 34.0] | -3.2 (14.9) [lower limit 14.9] | 41.4 (31.2) [lower limit 31.2]

68. Secondary Outcome: Percent Change From Baseline in IGF-1 at Week 54 - Females
Description: IGF-1 is a biochemical marker of growth hormone action and growth. The percent change from baseline in IGF-1 = ([IGF-1 value at Week 54] - [baseline IGF-1 value]) ÷ [baseline IGF-1 value] × 100.
Time Frame: Baseline and Week 54
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 30 | 42 | 4 | 1
Percent Change | -1.5 (34.4) | 7.2 (57.6) | -11.9 (13.4) | -13.5 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

69. Secondary Outcome: Percent Change From Baseline in IGF-1 at Week 20 - Males
Description: as for outcome 67
Time Frame: Baseline and Week 20
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 36 | 20 | 2 | 2
Percent Change | -2.7 (22.1) [lower limit 22.1] | 9.3 (29.6) [lower limit 29.6] | 7.6 (17.4) [lower limit 17.4] | 5.3 (16.2) [lower limit 16.2]

70. Secondary Outcome: Percent Change From Baseline in IGF-1 at Week 54 - Males
Description: as for outcome 68
Time Frame: Baseline and Week 54
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 32 | 18 | 1 | 2
Percent Change | -4.9 (33.5) | 29.6 (99.8) | 18.8 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed. | -6.8 (22.1)

71. Secondary Outcome: Percent Change From Baseline in Insulin-like Growth Factor Binding Protein 3 (IGF-BP3) at Week 20 - Females
Description: IGF-BP3 is a biochemical marker of growth hormone action and growth. The percent change from baseline in IGF-BP3 = ([IGF-BP3 value at Week 20] - [baseline IGF-BP3 value]) ÷ [baseline IGF-BP3 value] × 100.
Time Frame: Baseline and Week 20
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 41 | 50 | 6 | 2
Percent Change | 3.5 (18.2) [lower limit 18.2] | 3.8 (13.8) [lower limit 13.8] | 8.4 (12.9) [lower limit 12.9] | -0.7 (24.1) [lower limit 24.1]

72. Secondary Outcome: Percent Change From Baseline in IGF-BP3 at Week 54 - Females
Description: IGF-BP3 is a biochemical marker of growth hormone action and growth. The percent change from baseline in IGF-BP3 = ([IGF-BP3 value at Week 54] - [baseline IGF-BP3 value]) ÷ [baseline IGF-BP3 value] × 100.
Time Frame: Baseline and Week 54
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 31 | 45 | 4 | 2
Percent Change | 2.0 (16.7) | 4.5 (17.0) | 11.4 (17.4) | -13.4 (9.9)

73. Secondary Outcome: Percent Change From Baseline in IGF-BP3 at Week 20 - Males
Description: as for outcome 71
Time Frame: Baseline and Week 20
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 36 | 24 | 2 | 2
Percent Change | 5.6 (13.3) [lower limit 13.3] | 10.2 (18.6) [lower limit 18.6] | 3.3 (0.5) [lower limit 0.5] | 14.2 (50.6) [lower limit 50.6]

74. Secondary Outcome: Percent Change From Baseline in IGF-BP3 at Week 54 - Males
Description: as for outcome 72
Time Frame: Baseline and Week 54
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 32 | 21 | 1 | 2
Percent Change | 5.4 (18.4) | 18.2 (43.1) | -2.9 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed. | 22.5 (8.3)

75. Secondary Outcome: Growth Velocity at Week 20 - Females
Description: Growth Velocity (cm/year) = (Change from Baseline in height)/(Change from Baseline in chronologic age).
Time Frame: Week 20
Population: The analysis population included all female randomized participants who received ≥1 dose of study medication and had height data for the analysis endpoint at both baseline and Week 20.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 46 | 53 | 6 | 3
cm/year | 3.2 (8.2) [lower limit 8.2] | 1.9 (2.7) [lower limit 2.7] | 5.0 (6.8) [lower limit 6.8] | 0.6 (1.6) [lower limit 1.6]

76. Secondary Outcome: Growth Velocity at Week 54 - Females
Description: Growth Velocity (cm/year) = (Change from Baseline in height)/(Change from Baseline in chronologic age).
Time Frame: Week 54
Population: The analysis population included all female randomized participants who received ≥1 dose of study medication and had height data for the analysis endpoint at both baseline and Week 54.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 37 | 48 | 5 | 3
cm/year | 2.1 (3.7) | 1.2 (1.8) | 2.4 (2.9) | 0.7 (1.0)

77. Secondary Outcome: Growth Velocity at Week 20 - Males
Description: Growth Velocity (cm/year) = (Change from Baseline in height)/(Change from Baseline in chronologic age).
Time Frame: Week 20
Population: The analysis population included all male randomized participants who received ≥1 dose of study medication and had height data for the analysis endpoint at both baseline and Week 20.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 38 | 29 | 2 | 2
cm/year | 2.6 (2.7) [lower limit 2.7] | 3.6 (3.2) [lower limit 3.2] | -1.0 (1.3) [lower limit 1.3] | 1.7 (2.4) [lower limit 2.4]

78. Secondary Outcome: Growth Velocity at Week 54 - Males
Description: Growth Velocity (cm/year) = (Change from Baseline in height)/(Change from Baseline in chronologic age).
Time Frame: Week 54
Population: The analysis population included all male randomized participants who received ≥1 dose of study medication and had height data for the analysis endpoint at both baseline and Week 54.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 35 | 25 | 1 | 2
cm/year | 2.5 (2.5) | 2.8 (2.1) | 1.7 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed. | 2.8 (4.0)

79. Secondary Outcome: Skeletal Maturation at Week 20 - Females
Description: Skeletal Maturation = (Change from Baseline in bone age)/(Change from Baseline in chronologic age). Bone age was determined from an X-ray of left hand and wrist.
Time Frame: Week 20
Population: The analysis population included all female randomized participants who received ≥1 dose of study medication and had bone age data for the analysis endpoint at both baseline and Week 20.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 17 | 18 | 3 | 2
Ratio | 0.6 (1.9) [lower limit 1.9] | 0.4 (1.8) [lower limit 1.8] | 1.7 (2.3) [lower limit 2.3] | -0.8 (5.5) [lower limit 5.5]

80. Secondary Outcome: Skeletal Maturation at Week 54 - Females
Description: Skeletal Maturation = (Change from Baseline in bone age)/(Change from Baseline in chronologic age). Bone age was determined from X-ray of left hand and wrist. All participants in the Placebo/Sitagliptin arm were missing baseline or Week 54 measurements.
Time Frame: Week 54
Population: The analysis population included all female randomized participants who received ≥1 dose of study medication and had bone age data for the analysis endpoint at both baseline and Week 54.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 8 | 14 | 3 | 0
Ratio | 1.3 (1.1) | 1.0 (0.6) | 1.3 (2.2) |

81. Secondary Outcome: Skeletal Maturation at Week 20 - Males
Description: Skeletal Maturation = (Change from Baseline in bone age)/(Change from Baseline in chronologic age). Bone age was determined from X-ray of left hand and wrist.
Time Frame: Week 20
Population: The analysis population included all male randomized participants who received ≥1 dose of study medication and had bone age data for the analysis endpoint at both baseline and Week 20.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 13 | 17 | 1 | 1
Ratio | 1.6 (1.7) | 1.2 (1.1) | 0.4 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed. | 2.4 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed.

82. Secondary Outcome: Skeletal Maturation at Week 54 - Males
Description: Skeletal Maturation = (Change from Baseline in bone age)/(Change from Baseline in chronologic age). Bone age was determined from X-ray of left hand and wrist. All participants in the Metformin and Placebo/Sitagliptin arms were missing baseline or Week 54 measurements.
Time Frame: Week 54
Population: The analysis population included all male randomized participants who received ≥1 dose of study medication and had bone age data for the analysis endpoint at both baseline and Week 54.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 11 | 10 | 0 | 0
Ratio | 1.3 (0.9) | 1.3 (0.6) |  |

83. Secondary Outcome: Change From Baseline in Tanner Staging for Genitalia at Week 20 - Males
Description: Participant's stage of sexual maturation was assessed using the Tanner staging measure for determining pubertal development in male participants. Tanner staging includes an assessment of genital development (males) with a score of range 1 to 5 where 1=no development and 5=adult genitals. This change from baseline was Week 20 Tanner Staging for Genitalia minus the Week 0 Tanner Staging for Genitalia.
Time Frame: Baseline and Week 20
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 31 | 29 | 1 | 2
Score on a scale | 0.3 (0.5) | 0.2 (0.4) | 0.0 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed. | 0.5 (0.7)

84. Secondary Outcome: Change From Baseline in Tanner Staging for Genitalia at Week 54 - Males
Description: Participant's stage of sexual maturation was assessed using the Tanner staging measure for determining pubertal development in male participants. Tanner staging includes an assessment of genital development (males) with a score of range 1 to 5 where 1=no development and 5=adult genitals. This change from baseline was Week 54 Tanner Staging for Genitalia minus the Week 0 Tanner Staging for Genitalia. All participants in the Metformin arm were missing baseline or Week 54 measurements.
Time Frame: Baseline and Week 54
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 26 | 23 | 0 | 2
Score on a scale | 0.5 (0.6) | 0.6 (0.7) |  | 0.6 (0.7)

85. Secondary Outcome: Change From Baseline in Tanner Staging for Breasts at Week 20 - Females
Description: Participant's stage of sexual maturation was assessed using the Tanner staging measure for determining pubertal development in female participants. Tanner staging includes an assessment of breast development (females). Tanner stage (breast) is a score of range 1 to 5 where 1=no development and 5=adult breast. This change from baseline was Week 20 Tanner Staging for Breasts minus the Week 0 Tanner Staging for Breasts.
Time Frame: Baseline and Week 20
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 38 | 44 | 5 | 3
Score on a Scale | 0.2 (0.6) [lower limit 0.6] | 0.1 (0.3) [lower limit 0.3] | 0.2 (0.4) [lower limit 0.4] | 0.3 (0.6) [lower limit 0.6]

86. Secondary Outcome: Change From Baseline in Tanner Staging for Breasts at Week 54 - Females
Description: Participant's stage of sexual maturation was assessed using the Tanner staging measure for determining pubertal development in female participants. Tanner staging includes an assessment of breast development (females). Tanner stage (breast) is a score of range 1 to 5 where 1=no development and 5=adult breast. This change from baseline was Week 54 Tanner Staging for Breasts minus the Week 0 Tanner Staging for Breasts.
Time Frame: Baseline and Week 54
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 28 | 36 | 4 | 3
Score on a Scale | 0.5 (0.7) | 0.4 (0.6) | 0.5 (1.0) | 0.7 (0.6)

87. Secondary Outcome: Change From Baseline in Tanner Stage for Pubic Hair at Week 20 - Females
Description: Participant's stage of sexual maturation was assessed using the Tanner staging measure for determining pubertal development in female participants. Tanner staging includes an assessment of pubic hair development (females). Tanner stage (pubic hair) is a score of range 1 to 5 where 1=no development and 5=adult pubic hair. This change from baseline was Week 20 Tanner Staging for Pubic Hair minus the Week 0 Tanner Staging for Pubic Hair.
Time Frame: Baseline and Week 20
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 38 | 43 | 5 | 3
Score on a scale | 0.1 (0.4) [lower limit 0.4] | 0.1 (0.3) [lower limit 0.3] | 0.2 (0.4) [lower limit 0.4] | 0.0 (0.0) [lower limit 0.0]

88. Secondary Outcome: Change From Baseline in Tanner Stage for Pubic Hair at Week 54 - Females
Description: Participant's stage of sexual maturation was assessed using the Tanner staging measure for determining pubertal development in female participants. Tanner staging includes an assessment of pubic hair development (females). Tanner stage (pubic hair) is a score of range 1 to 5 where 1=no development and 5=adult pubic hair. This change from baseline was Week 54 Tanner Staging for Pubic Hair minus the Week 0 Tanner Staging for Pubic Hair.
Time Frame: Baseline and Week 54
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 28 | 35 | 4 | 3
Score on a scale | 0.5 (0.6) | 0.3 (0.5) | 0.8 (1.5) | 0.3 (0.6)

89. Secondary Outcome: Change From Baseline in Tanner Stage for Pubic Hair at Week 20 - Males
Description: Participant's stage of sexual maturation was assessed using the Tanner staging measure for determining pubertal development in male participants. Tanner staging includes an assessment of pubic hair development (males). Tanner stage (pubic hair) is a score of range 1 to 5 where 1=no development and 5=adult pubic hair. This change from baseline was Week 20 Tanner Staging for Pubic Hair minus the Week 0 Tanner Staging for Pubic Hair.
Time Frame: Baseline and Week 20
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 32 | 29 | 1 | 2
Score on a scale | 0.3 (0.5) | 0.2 (0.4) | 0.0 (NA) — "NA" The standard deviation could not be calculated because only one participant was analyzed. | 0.5 (0.7)

90. Secondary Outcome: Change From Baseline in Tanner Stage for Pubic Hair at Week 54 - Males
Description: Participant's stage of sexual maturation was assessed using the Tanner staging measure for determining pubertal development in male participants. Tanner staging includes an assessment of pubic hair development (males). Tanner stage (pubic hair) is a score of range 1 to 5 where 1=no development and 5=adult pubic hair. This change from baseline was Week 54 Tanner Staging for Pubic Hair minus the Week 0 Tanner Staging for Pubic Hair.
Time Frame: Baseline and Week 54
Population: The analysis population included all male randomized participants who received ≥1 dose of study medication and had data for the analysis endpoint at both baseline and Week 54. Tanner staging results for pubic hair were unavailable for the Metformin arm.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 26 | 23 | 0 | 2
Score on a scale | 0.5 (0.7) | 0.6 (0.5) |  | 0.5 (0.7)

91. Secondary Outcome: Participants With Worsening in Dental Status at Week 20
Description: Participants were evaluated with a visual oral exam; a subset had dental photographs. Teeth worsening was defined as worsening of tooth fracture, tooth discoloration, or enamel defect as determined by an independent reviewer. Worsening in these categories was a change in dental defect assessments made by comparing Week 20 dental assessments versus baseline dental assessments.
Time Frame: Week 20
Population: The analysis population included all randomized participants who received ≥1 dose of study medication and had dental data at baseline and Week 20.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 88 | 85 | 8 | 5
Participants
  1. With ≥1 tooth with worsening in any category | 32 | 25 | 1 | 0
  2. With ≥1 tooth with worsening fracture | 5 | 5 | 0 | 0
  3. With ≥1 tooth with worsening discoloration | 29 | 23 | 0 | 0
  4. With ≥1 tooth with worsening enamel defect | 7 | 4 | 1 | 0

92. Secondary Outcome: Participants With Worsening in Dental Status at Week 54
Description: Participants were evaluated with a visual oral exam; a subset had dental photographs. Teeth worsening was defined as worsening of tooth fracture, tooth discoloration, or enamel defect as determined by an independent reviewer. Worsening in these categories was a change in dental defect assessments made by comparing Week 54 dental assessments versus baseline dental assessments.
Time Frame: Week 54
Population: The analysis population included all randomized participants who received ≥1 dose of study medication and had dental data at baseline and Week 54.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
Number analyzed (Participants) | 79 | 78 | 8 | 5
Participants
  1. With ≥1 tooth with worsening in any category | 49 | 50 | 2 | 0
  2. With ≥1 tooth with worsening fracture | 13 | 15 | 1 | 0
  3. With ≥1 tooth with worsening discoloration | 45 | 48 | 2 | 0
  4. With ≥1 with worsening enamel defect | 13 | 13 | 1 | 0

ADVERSE EVENTS:
Time Frame: SAEs and AEs: Up to approximately Week 56. Deaths: Up to approximately 42 months after randomization.
Description: The All-Cause Mortality analysis population consisted of all randomized participants. The AE analysis population consisted of all participants who received ≥1 dose of study medication and included all post-randomization follow-ups. One participant in the Sitagliptin arm died after the treatment phases of the study, approximately 42 months after randomization.
Arm/Group | Sitagliptin | Placebo/Metformin | Metformin | Placebo/Sitagliptin
All-Cause Mortality (participants affected / at risk) | 1/96 | 0/90 | 0/9 | 0/5
Serious Adverse Events (participants affected / at risk) | 10/95 | 7/90 | 1/9 | 3/5
Other Adverse Events (participants affected / at risk) | 62/95 | 53/90 | 7/9 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=95) | Placebo/Metformin (N=90) | Metformin (N=9) | Placebo/Sitagliptin (N=5)
Gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abscess soft tissue (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sexual abuse (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=95) | Placebo/Metformin (N=90) | Metformin (N=9) | Placebo/Sitagliptin (N=5)
Wandering pacemaker (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 8 (10) | 7 (10) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 11 (14) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (6) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (5) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (9) | 7 (8) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 6 (7) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (4) | 7 (10) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 6 (7) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 15 (19) | 6 (6) | 0 (0) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 6 (7) | 6 (6) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 12 (15) | 12 (13) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 9 (11) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 3 (3) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 16 (107) | 12 (37) | 3 (65) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 3 (5) | 2 (2) | 0 (0) | 2 (4)
Headache (Nervous system disorders) | 9 (9) | 13 (16) | 2 (5) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 1 (2) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/ presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT01485614/Prot_SAP_000.pdf